CLINICAL TRIAL: NCT00906217
Title: Safety, Efficacy, and Tolerance of Pico-Salax for Colon Cleansing Prior to Colonoscopy in an Elderly Population
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Lawrence Charles Hookey, assistant professor of medicine, Queen's University
Other Study IDs: Hookey Picosalax Elderly Trial
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Colon Cleansing
Keywords: colonoscopy; preparation; safety; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elderly patients: patients older than 70 years with normal renal function

SUMMARY:
This study aims to further define the appropriate population for Pico-Salax, a purgative used prior to colonoscopy. Patients over the age of 70 years with normal renal function scheduled for colonoscopy will receive Pico-Salax and have pre and post preparation bloodwork and electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

* >70 years

Exclusion Criteria:

* renal dysfunction
* congestive heart failure
* ileus

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients older than 70 scheduled for colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
serum electrolyte changes pre and post preparation | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Principal Investigator — Queen's University